CLINICAL TRIAL: NCT01710072
Title: Aspirin as a Promising Agent to Attenuate Inflammation in the Wall of Human Cerebral Aneurysms
Brief Title: Aspirin Attenuates Inflammation in Human Cerebral Aneurysms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, David Hasan, Assistant Professor and Section Chief, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 201108750
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: The Focus of the Study is to Monitor MRI Signal Changes and Inflammatory Biomarkers With Use of Aspirin in Patients With Unruptured Cerebral Aneurysm
Keywords: aneurysm, inflammation, MRI
MeSH Terms: conditions — Aneurysm; Inflammation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Experimental): aspirin 81 mg po every day
  Interventions: Drug: aspirin
- no aspirin (No Intervention)

INTERVENTIONS:
Drug: aspirin
  Arms: aspirin

SUMMARY:
Hypothesis: aspirin attenuates inflammation in cerebral aneurysms and hence reduces the incidence of rupture. This effect can be monitored using the signal generated by macrophages (inflammatory biomarker) in ferumoxytol-enhanced MRI.

Study aims:

1. Determine if daily aspirin intake (for three months) would obliterate/reduce ferumoxytol-enhanced MRI signal changes generated by macrophages in cerebral aneurysm wall. Fifteen patients with cerebral aneurysms > 7 mm will be selected to enroll in this pilot study. 10 patients will be imaged at base line with ferumoxytol-enhanced MRI. Following that, they will take aspirin 81 mg daily and then re-imaged again at three months. This group will be compared to a control group of 5 patients where they will have the imagings studies performed at base line and at three months but will NOT take aspirin.

DETAILED DESCRIPTION:
If you are eligible to enroll in the study, you will be contacted by the principal investigator in person and he will describe the study in a private setting (neurosurgery clinic room or hospital patient room). You will be given ample opportunity to decide to participate or not.

You will be randomly assigned to receive one of the 2 study treatments, either taking aspirin or not. This means that whichever study treatment you receive will be determined purely by chance, like flipping a coin. You will have a 2 out of 3 chance of receiving the study treatment (aspirin). You will be told which study treatment arm you are on.

A 15 minute base line MRI of the brain will be performed initially. Following that, the medication (ferumoxytol) will be injected intravenously over 3 minutes. The second MRI of the brian will obtained 24 hours later. A third MRI will be obtained also at 72 hours following the injection of medication. Then after the third MRI, ten people will be chosen randomly to start aspirin every day for three months total. The selected aspirin group will be given 3-month supply of aspirin (81 mg). The other five patients will be asked to avoid any anti-inflammatory drugs (like aspirin, Advil, ibuprofen, …) if at all possible. Following an interval of three months, a repeat MRI of the brain will be done exactly as above (a base line MRI of the brain will be done, then the medication will be injected intravenously (IV). A second MRI will be obtained 24 hours later followed by another one at 72 hours later.

MRI scans:

An MRI scanner takes pictures of the inside of your brain. You will be asked to lie on your back on a special table that slides into the tube. The sides of the tube will be fairly close to your body and the scanner makes a loud hammering noise while you are inside. You will be able to talk to people in the room through a speaker system. We will monitor you closely while you are inside the scanner.

The MRI images for this study are not being used to evaluate your health. The images obtained for this study are for specific research purposes and are not being used to find medical abnormalities. These images will not be reviewed by a radiology physician to diagnose existing abnormalities.

Sequence of events:

1. Informed consent will be obtained.
2. Serum pregnancy test (if you are a female of child bearing age) and blood chemistry labs will be collected. If the results are positive, you will not be able to continue in the study.
3. IV access will be inserted.
4. 15-30 minutes base-line MRI will be performed
5. The study medication, ferumoxytol, will be given to you via IV line immediately after the first MRI
6. The second MRI will be obtained 24 hours later
7. The third MRI will be obtained 72 hours following infusion of ferumoxytol.
8. You will be selected randomly to either receive aspirin or not.
9. Ten patients will be assigned to start taking aspirin (325mg) every day for 3 months.
10. Five patients will be asked to avoid any anti-inflammatory drugs (like aspirin, Advil, ibuprofen…) for three months if all possible.
11. At three months, another base-line MRI will be performed
12. The study medication, ferumoxytol, will be given to you via IV line immediately after the first MRI
13. The second MRI will be obtained 24 hours later
14. The third MRI will be obtained 72 hours following infusion of ferumoxytol
15. Study is finished

WHAT ARE THE RISKS OF THIS STUDY? What are the risks of the study? You may experience one or more of the risks indicated below from being in this study. In addition to these, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study.

Aspirin:

1. Nausea 2. Vomiting 3. Stomachache/burn 3 Stomach pain suggestive of stomach ulcer 5. Black stool suggestive of rectal bleeding 6. Dizziness 7. Rash 8. Fever

Ferumoxytol:

1. Diarrhea (4%),
2. nausea (3.1%),
3. dizziness (2.6%),
4. hypotension (2.5%),
5. constipation (2.1%),
6. swelling of the legs, arms and/or face (2%),
7. headache (1.8%),
8. edema (1.5%),
9. vomiting (1.5%),
10. abdominal pain (1.3%),
11. chest pain (1.3%),
12. cough (1.3%),
13. rash (1%),
14. muscle spasm (1%),
15. back pain (1%),
16. hypertension (1%),
17. shortness of breath (1%),
18. itching (1%).
19. life-threatening or severe allergic reaction that could lead to death

MRI Scan:

You may be uncomfortable inside the MRI scanner if you do not like to be in closed spaces ("claustrophobia"). During the procedure, you will be able to talk with the MRI staff through a speaker system. You can tell them to stop the scan at any time.

The MRI produces a loud hammering noise, which has produced hearing loss in a very small number of patients. You will be given earplugs to reduce this risk.

Loss of confidentiality:

1. your name, diagnosis, age, gender and potential treatment could be accessed by non-research team individuals.

Intravenous Catheter Insertion:

For this study you will need to have small amount of blood drawn for laboratory studies to make sure that it is safe for you to participate in the study. You will have an intravenous catheter (IV) placed peripherally (usually arm or hand) for infusion of the study drug, ferumoxytol. There are minimal risks associated with placement of the IV, including pain, bleeding, bruising, and infection at the IV site.

Women Capable of Becoming Pregnant If you are a woman who is capable of becoming pregnant, we will ask you to have a pregnancy test before beginning this study. You must use effective birth control methods and try not to become pregnant while participating in this study. If you become pregnant, there may be unknown risks to your fetus, or risks to your fetus that we did not anticipate, associated with being in the study. There may be long-term effects of the treatment being studied that could increase the risk of harm to an unborn child. If you believe or know you have become pregnant while participating in this research study, please contact David Hasan 319-384-8669 as soon as possible.

WHAT ARE THE BENEFITS OF THIS STUDY? You will not benefit from being in this study.

However, we hope that, in the future, other people might benefit from this study because it may inform us if taking aspirin daily would help stabilize the aneurysm wall and reduce the risk of rupture.

WHAT OTHER TREATMENT OPTIONS ARE THERE?

Before you decide whether or not to be in this study, your doctor will discuss the other options that are available to you. Instead of being in this study, you could undergo microsurgical clipping of your aneurysm, have your aneurysm treated endovascularly by placing coils in the aneurysm sac, or just observe your aneurysm and monitored with imaging studies.

WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

You will not have any additional costs for being in this research study. All the costs associated with MRIs and the injections will be covered by the study. There may be additional costs associated with travel to and from visits.

You and/or your medical/hospital insurance carrier will remain responsible for your regular medical care expenses.

WILL I BE PAID FOR PARTICIPATING?

You will not be given any direct compensation for being in this research study. However, the study will pay for any hotel accommodation that may be given should you need lodging between MRI visits.

WHO IS FUNDING THIS STUDY?

The University and the research team are receiving no payments from other agencies, organizations, or companies to conduct this research study.

WHAT IF I AM INJURED AS A RESULT OF THIS STUDY?

* If you are injured or become ill from taking part in this study, medical treatment is available at the University of Iowa Hospitals and Clinics.
* The University of Iowa does not plan to provide free medical care or payment for treatment of any illness or injury resulting from this study unless it is the direct result of proven negligence by a University employee.
* If you experience a research-related illness or injury, you and/or your medical or hospital insurance carrier will be responsible for the cost of treatment.

WHAT ABOUT CONFIDENTIALITY? We will keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people such as those indicated below may become aware of your participation in this study and may inspect and copy records pertaining to this research. Some of these records could contain information that personally identifies you.

* federal government regulatory agencies,
* the U.S. Food and Drug Administration
* auditing departments of the University of Iowa, and
* the University of Iowa Institutional Review Board (a committee that reviews and approves research studies)

To help protect your confidentiality, you will not be identified by name, social security number, address or phone number. The hard copy and electronic records will include a code number and initials. The list that matches your name with the code number will be kept in password protected computer file in Dr. Hasan's locked office. Also the hard copies of your study material will be kept in locked file cabinets in a locked office. If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

The University of Iowa Hospitals and Clinics generally requires that we document in your medical record chart that you are participating in this study. The information included in the chart will provide contact information for the research team as well as information about the risks associated with this study. We will keep this Informed Consent Document in our research files; it will not be placed in your medical record chart.

IS BEING IN THIS STUDY VOLUNTARY?

Taking part in this research study is completely voluntary. You may choose not to take part at all. If you decide to be in this study, you may stop participating at any time. If you decide not to be in this study, or if you stop participating at any time, you won't be penalized or lose any benefits for which you otherwise qualify.

What if I Decide to Drop Out of the Study?

If you decided to drop out of the study, you will not suffer any adverse consequences (physical, social, economic, legal or psychological).

Will I Receive New Information About the Study while Participating? If we obtain any new information during this study that might affect your willingness to continue participating in the study, we'll promptly provide you with that information.

Can Someone Else End my Participation in this Study? Under certain circumstances, the researchers might decide to end your participation in this research study earlier than planned. This might happen if your aneurysm ruptures or becomes symptomatic.

WHAT IF I HAVE QUESTIONS?

We encourage you to ask questions. If you have any questions about the research study itself, please contact: David Hasan, MD, 319-331-1459. If you experience a research-related injury, please contact:

David Hasan MD, 319-331-1459.

If you have questions, concerns, or complaints about your rights as a research subject or about research related injury, please contact the Human Subjects Office, 105 Hardin Library for the Health Sciences, 600 Newton Rd, The University of Iowa, Iowa City, IA 52242-1098, (319) 335-6564, or e-mail irb@uiowa.edu. General information about being a research subject can be found by clicking "Info for Public" on the Human Subjects Office web site, http://research.uiowa.edu/hso. To offer input about your experiences as a research subject or to speak to someone other than the research staff, call the Human Subjects Office at the number above.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years.
2. Incidental (non-ruptured) IA ≥5 mm.
3. Treating neurosurgeon and patient agree on observation period of 3 months before proceeding with treatment either endovascularly or by microsurgical clipping.
4. Positive MRI signal change corresponding of ferumoxytol uptake is observed.
5. No history of aspirin intake or NSAIDs for 4 weeks prior to enrolment.
6. No current history of statin use.

Exclusion Criteria:

1. Patients with treated IAs (by coil embolization or surgical clipping) will be excluded.
2. Patients presenting with ruptured intracranial IAs will also be excluded from the study, to avoid interfering with timely treatment of ruptured IAs.
3. Children
4. pregnant women
5. persons with history of allergy or hypersensitivity to iron or dextran or iron-polysaccharide preparations
6. patients requiring monitored anesthesia or intravenous (IV) sedation for MR imaging
7. patients with contraindication to MRI
8. patients with renal insufficiency, hepatic insufficiency or iron overload, 9. patients receiving combination antiretroviral therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
measurement of inflammatory biomarkers | 3 months
  At the end of treatment, Inflammatory biomarkers are used to assess the efficacy of treatment (aspirin)

SECONDARY OUTCOMES:
change in the signal intensity of MRI | 3 months
  at the end of the 3 months, the MRI signal intensity are measured and compared to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Hasan DM, Chalouhi N, Jabbour P, Dumont AS, Kung DK, Magnotta VA, Young WL, Hashimoto T, Richard Winn H, Heistad D. Evidence that acetylsalicylic acid attenuates inflammation in the walls of human cerebral aneurysms: preliminary results. J Am Heart Assoc. 2013 Feb 22;2(1):e000019. doi: 10.1161/JAHA.112.000019. PMID 23525414